CLINICAL TRIAL: NCT01692106
Title: A Clinical Study of Per Oral Endoscopic Myotomy (POEM) in Patients Suffering From Achalasia.
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Dennis Hong MD, Dr. Dennis Hong, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2012-09-19; First posted 2012-09-25 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Achalasia
Keywords: Heller myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peroral endoscopic myotomy (POEM) (Experimental): The Procedure: per oral endoscopic myotomy (POEM)will be performed on all patients in this single arm study.
  Interventions: Procedure: Procedure: Per Oral Endoscopic Myotomy (POEM)

INTERVENTIONS:
Procedure: Procedure: Per Oral Endoscopic Myotomy (POEM) — lower esophageal sphincter muscle is sectioned through an unique endoscopic approach.

SUMMARY:
This study evaluates the feasibility of endoscopic myotomy for achalasia. In achalasia, there is loss of relaxation of the lower esophageal sphincter (LES), as well as a higher baseline pressure in the LES. The most widespread treatment for this disease and the one that has the best long term results involves cutting the muscle layers of the lower esophagus and on the neighbouring stomach without injurying the underlying mucosa or inner layer of the esophageal wall. This is done during a surgery through the abdomen either with a big incision or more recently with the keyhole technique. This surgery has various potential complications, one of which being making a hole through the mucosa or not extending the cut on the muscle long enough to obtain adequate relaxation of the sphincter. The per oral endoscopic myotomy (POEM) is a new intervention that is done also under general anesthesia in the operating room; however, it involves no skin incisions and all the procedure is done through a fiber optic camera. It involves making a cut in the inner layer of the esophagus and then with cautery cut the muscle fibers responsible of the blockage and finally closing the initial opening with clips. In this study we will investigate the feasibility of this intervention both from a technical aspect as well as a logistical perspective given the local operating room constraints.

DETAILED DESCRIPTION:
All patients will have routine pre-operative EGD, manometry, barium swallow, ph-metry. Equally all patients will undergo Eckardt's and grading systems of symptom severity before and after the intervention. The patients will have a gastro-graffin swallow in the first day after the surgery.

Procedure: Under general anesthesia upper endoscopy is performed using a standard single channel gastroscope. Submucosal injection with 10 ml saline with 1% methylen blue at the level of the mid esophagus is initially performed. A small longitudinal submucosal incision is created using a standard needle knife. For a sufficient entry point as well as submucosal tunnel, a dilating balloon is inserted submucosally via the created incision similar to the technique used in standard endoscopic submucosal dissection. The balloon is slightly inflated to allow sufficient entrance of the endoscope. The gastroscope is advanced into the submucosal space and the tunnel is created via needle knife or blunt dissection as appropriate. The tunnel is created distally and is stopped several centimeters beyond the lower esophageal sphincter (LES), which can easily be identified. Using flexible scissors, a triangle tip- or respectively an isolated tip-knife the clearly visible circular muscles are divided starting 4 cm above the LES extending 2 cm beyond the previously identified esophageal border. The longitudinal and serosal layers are left intact. Finally the mucosal entry is closed with standard endoscopic clips. Patients will receive standard postoperative care for surgical myotomy, including long-term follow-up.

If for any reason the endoscopic treatment is unable to be completed or infeasible, a standard laparoscopic treatment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for a Heller myotomy
* No contra-indication to general anesthesia
* Their age is ≥18 years and ≤80 years
* Able to give written consent

Exclusion Criteria:

* Previous intervention for achalasia: any of previous Heller myotomy, Botox injections, endoscopic myotomy
* Previous mediastinal surgery
* Any anatomical esophageal anomaly that in the opinion of the investigator may render the intervention more difficult, such as sigmoid esophagus on the pre-operative barium swallow or hiatal hernia > 2cm.
* Body mass index (BMI) > 40
* Any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
feasibility of the POEM procedure in achalasia | 1-6 months
  Patients will be consecutively evaluated on effectiveness of the endoluminal procedure by conducting standard diagnostics including postoperative gastrografin swallow. After 6 months standard esophagogastroduodenoscopy (EGD), high-resolution manometry and pH impedance will be done and a Quality of Life questionnaire will be filled out. Results will be compared to historical data of 40 conventional laparoscopic Heller myotomies.

SECONDARY OUTCOMES:
complications | 1-6 months
  post-operative complications, intra-operative outcomes as well as the Eckardt's grading systems of symptom severity and reflux grading secondary to achalasia.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD, Principal Investigator — St. Josephs' Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada